CLINICAL TRIAL: NCT02765945
Title: The Effect of Long-term Exercise on the Production of Osteoclastogenic and Anti-osteoclastogenic Cytokines by Peripheral Blood Mononuclear Cells and on Serum Markers of Bone Metabolism
Brief Title: Exercise as an Modulator of Immunological Risk Factors for Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Tennessee State University (Other)
Responsible Party: Principal Investigator, John Kelly Smith, Emeritus Professor of Medicine, East Tennessee State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 96-028f
Record Dates: First submitted 2016-05-05; First posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Osteoporosis
Keywords: Exercise; Osteoporosis; Cytokines
MeSH Terms: conditions — Osteoporosis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Supervised exercise program — Subjects were enrolled in a hospital-based wellness center where, after analysis of their medical history and previous levels of physical activity ands documentation of a normal exercise stress test, they chose individually tailored exercise programs

SUMMARY:
This is the second phase of a study designed to determine the immunological effects of long-term exercise on risk factors for ischemic heart disease (phase 1) and osteoporosis (phase 2). The results indicate that six months of moderate intensity exercise reduces bone resorption and increases the secretion of anti-osteoclastogenic cytokines by peripheral blood mononuclear cells.

DETAILED DESCRIPTION:
In a before and after trial involving 43 healthy adults the investigators measured the effect of six months of supervised exercise on the spontaneous and phytohemagglutinin-induced production of osteoclastogenic cytokines (interleukin-1α, tumor necrosis factor-α), anti-osteoclastogenic cytokines (transforming growth factor-β, interleukins 4 and10), pleiotropic cytokines with variable effects on osteoclastogenesis (interferon-γ, interleukin-6), and T cell growth and differentiation factors (interleukins 2 and 12) by peripheral blood mononuclear cells. The investigators also measured lymphocyte phenotypes, and serum markers of bone formation (osteocalcin), bone resorption (C-terminal telopeptides of Type I collagen), and bone homeostasis (estradiol, vitamin D2, testosterone, parathyroid hormone, insulin-like growth factor).

ELIGIBILITY:
Inclusion Criteria:

* Normal exercise treadmill test

Exclusion Criteria:

* Any medical condition that would prevent participation in a six month exercise program

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 1996-12; Primary Completion 1998-04 (Actual); Study Completion 1998-04 (Actual)

PRIMARY OUTCOMES:
Evidence of altered bone resorption and/or production as measured by measurements of serum levels of osteocalcin and degradation products of Type I collagen (C-terminal telopeptides) | 6 months
Evidence of altered secretion of osteoclastogenic cytokines by peripheral blood mononuclear cells | 6 months
  secretion of IL-1 alpha, TNF-alpha, IFN-gamma by cultured peripheral blood mononuclear cells
Evidence of altered secretion of anti-osteoclastogenic cytokines by cultured peripheral blood mononuclear cells | 6 months
  secretion of IL-10, IL-4, TGF-beta, IL-6 by cultured peripheral blood mononuclear cells
Evidence of altered blood mononuclear cell phenotypes | 6 months
  Immunophenotyping of blood mononuclear cells by FACScan flow cytometer
Evidence of altered serum factors of bone homeostasis | 6 months
  Measurements of serum levels of estradiol, testosterone, PTH, IGF-1
Evidence of altered secretion of growth and differentiation factors by cultures peripheral blood mononuclear cells | 6 months
  Measurements of IL-2, IL-4, IL-12

CONTACTS AND LOCATIONS:
Overall Officials: John K Smith, MD, Principal Investigator — James H. Quillen College of Medicine, Johnson City, Tennesse, United States 70571
Locations (1):
- James H. Quillen College of Medicine, Johnson City, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith JK, Dykes R, Chi DS. The Effect of Long-Term Exercise on the Production of Osteoclastogenic and Antiosteoclastogenic Cytokines by Peripheral Blood Mononuclear Cells and on Serum Markers of Bone Metabolism. J Osteoporos. 2016;2016:5925380. doi: 10.1155/2016/5925380. Epub 2016 Aug 24. PMID 27642534